#### NCT02087085

**Study ID:** 190342-038

**Title:** Safety and Efficacy of Brimonidine Posterior Segment Drug Delivery System in Patients with Geographic Atrophy Secondary to Age-related Macular Degeneration

Statistical Analysis Plan Date: 03-Aug-2018

#### 1. Title Page

#### STATISTICAL ANALYSIS PLAN

Safety and Efficacy of Brimonidine Posterior Segment Drug Delivery System in Patients with Geographic Atrophy Secondary to Age-Related Macular Degeneration (BEACON Study: 190342-038)

Version 2.0: 2018-08-03

Protocol Number: 190342-038 Amendment 7

Development Phase: 2b

Product Name: AGN-190342, Brimonidine Drug Delivery System

(Brimo DDS<sup>®</sup>)

Study Statistician:

Sponsor: Allergan (North America)

2525 Dupont Drive Irvine, California USA

92612

+1-714-246-4500 +1-800-347-4500

Allergan Ltd. 1st Floor, Marlow International,

The Parkway, Marlow Buckinghamshire

SL7 1YL United Kingdom Tel: +44 (0) 1628 494444 Fax: +44 (0) 1628 494449

This document is the property of Allergan, plc. and may not, in full or part, be passed on, reproduced, published, distributed to any person, or submitted to any regulatory authority without the express written permission of Allergan, plc.

| 2. | <b>Table of Contents</b> |
|----|--------------------------|
| 1. | Title Page |

| 1. | Title | e Page | 1 |
|---|---|---|---|
| 2. | Tabl | le of Contents | 2 |
| | 2.1 | List of Tables | 3 |
| | 2.2 | List of Figures | |
| 3. | | of Abbreviations and Definition of Terms | |
| 4. | | oduction | |
| | 4.1 | Study Design Summary | |
| | | 4.1.1 Overall Design | |
| | | 4.1.2 Number of Participants | |
| | 4.2 | Study Objectives and Endpoints | 8 |
| | 4.3 | Schedule of Activities | 9 |
| 5. | Stati | istical Methodology and Study Endpoints | 12 |
| | 5.1 | Statistical Methods Planned in the Protocol and Determination of Sample Size | 12 |
| | | 5.1.1 Statistical and Analytical Plans | 12 |
| | | 5.1.1.1 Common Conventions | 12 |
| | | 5.1.1.2 Demographics | 14 |
| | | 5.1.1.3 Efficacy Analyses | 16 |
| | | 5.1.1.5 Subgroup Analyses | 23 |
| | | 5.1.1.6 Interim Analyses | |
| | | 5.1.2 Determination of Sample Size | 23 |
| | 5.2 | Changes in the Conduct of the Study or Planned Analyses | 24 |
| | | 5.2.1 Changes in the Conduct of the Study | 24 |
| | | 5.2.2 Changes to Analyses Prior to Database Lock | 24 |
| 6. | Data | a Handling and Analysis Conventions | 25 |
| | 6.1 | Study Treatment Conventions. | 25 |
| | | 6.1.1 Analysis Days | 25 |
| | | 6.1.2 Missing/Incomplete Treatment End Date | 25 |
| | 6.3 | Site Pooling | |
| | 6.4 | Missing/Incomplete Date Conventions | 2 <i>e</i> |

| | 6.4.1 Missing/Incomplete Adverse Event (AE), Start Date | 27 |
|---|---|---|
| | 6.4.2 Missing/Incomplete Medication Start Date | |
| | 6.4.3 Missing/Incomplete AE/Medication End Date | |
| 6.5 | Efficacy Endpoint Conventions | |
| 6.6 | Safety Endpoint Conventions | 28 |
| | 6.6.1 Adverse Events | 28 |
| | 6.6.1.1 Missing Intensity or Relationship | |
| | 6.6.2 Repeated or Unscheduled Assessments of Safety Parameters | |
| 6.7 | Imputed Value Listing Conventions | |
| 6.8 | Handling Mis-randomization and Mis-stratification | 29 |
| 7. Refe | erences | |
| , 1010 | | |
| 2.1 | List of Tables | |
| Table 3- | Abbreviations and Definitions of Terms | 5 |
| Table 5- | 1 Analysis Populations | 12 |
| Table 5-2 | J I | |
| Table 5- | $\omega$ | |
| Table 5-4 | 4 Participant Disposition Summaries | 14 |
| Table 5- | 5 Protocol Deviation Summary | 15 |
| Table 5- | <b>U</b> 1 | |
| Table 5- | | |
| Table 5- | | |
| Table 5-9<br>Table 5- | | |
| Table 5- | | |
| Table 5- | 1 | |
| Table 5- | | |
| Table 5- | 1 3 | |
| Table 5- | AE Terms | 20 |
| Table 5- | | 20 |
| Table 5-2 | 27 Sample Size Assumption | 24 |

| Table 6-1 | Analysis Day Definitions | 25 |
|-----------|-------------------------------------------------------------|----|
| Table 6-4 | Imputation Scenarios | 26 |
| Table 6-5 | Initial Imputed Date Algorithm | 27 |
| Table 6-6 | Treatment Group Label in TFL | 27 |
| Table 6-7 | Programming Conventions | 28 |
| Table 6-8 | Missing AE Intensity and Relationship Imputation Algorithms | 28 |

# 2.2 List of Figures

No table of figures entries found.

# 3. List of Abbreviations and Definition of Terms

Table 3-1 Abbreviations and Definitions of Terms

| Abbreviation/Term | Definition |
|-------------------|----------------------------------------------|
| ACT | anatomical therapeutic chemical |
| AE | adverse event |
| AMD | age-related macular degeneration |
| BCVA | Best-corrected visual acuity |
| Brimo DDS® | Brimonidine Drug Delivery System |
| CRC | central reading center |
| cSLO | confocal scanning laser Ophthalmoscopy |
| eCRF | electronic case report form |
| ECG | electrocardiogram |
| Led | olectrocardiogram |
| ETDRS | early treatment diabetic retinopathy study |
| FAF | fundus autofluorescence |
| GA | geographic atrophy |
| | geograpme anophy |
| IOP | intraocular pressure |
| IR | infrared reflectance |
| IVRS | interactive voice response system |
| IWRS | interactive web response system |
| LLT | lowest level term |
| LOCF | last observation carried forward |
| MedDRA | medical dictionary for regulatory activities |
| mITT | modified intent-to-treat |
| MMRM | mixed-effects model for repeated measures |
| NA | non applicable |
| OC | observed cases |
| OCT | optical coherence tomography |
| OD | oculus dexter (the right eye) |
| OS | oculus sinister (the left eye) |
| OU | oculus uterque (both eyes) |
| PCS | potentially clinically significant |
| PID | patient identification |
| PP | per-protocol |
| PRO | patient-reported outcome |
| PT | preferred term |
| qFAF | quantitative fundus autofluorescence |
| SAE | serious adverse event |

| Abbreviation/Term | Definition |
|---|---|
| SAP | statistical analysis plan |
| SD-OCT | spectral-domain optical coherence tomography |
| SI | Le Système International d'Unités (International System of Units) |
| SOC | system organ class |
| TEAE | treatment-emergent adverse event |
| WHO DDE | the World Health Organization drug dictionary enhanced |

#### 4. Introduction

This statistical analysis plan (SAP) details comprehensive, technical specifications of the statistical analyses of the efficacy and safety data outlined and/or specified in the final protocol of Study 190342-038 (BEACON) and the most recent amendment (version 7). Specifications of tables, figures, and data listings are contained in a separate document. The SAP for microperimetry fundus autofluorescence (FAF) signal intensity, pharmacokinetic/pharmacodynamics (Blood samples for PK), genomic analysis (Blood Samples for Genotypic Analysis and Gene Expression Analysis) and health economics and health outcomes research data separately.

This document is organized into 3 main sections:

- 1. Study overview
- 2. Statistical Methodology and Study Endpoints
- 3. Data Handling and Analysis Conventions

#### 4.1 Study Design Summary

#### 4.1.1 Overall Design

This is a multicenter, double-masked, randomized, Sham treatment-controlled, 30-month phase 2b study designed to evaluate the safety and efficacy of Brimo DDS in patients with geographic atrophy (GA) secondary to age-related macular degeneration (AMD). Patients will be randomized in a 1:1 ratio to receive 400  $\mu$ g Brimo DDS, administered by intravitreal injection, or Sham treatment (control). Randomization will be stratified by region (North America, Europe, and Australia) and by atrophic lesion area ( $\leq 8 \text{ mm}^2 \text{ versus} > 8 \text{ mm}^2$ ) in the study eye as assessed by FAF examination at Screening Visit 1 and quantified by the Central Reading Center (CRC). The study medication will be administered every 3 months from Baseline (Day 1) through Month 21.

The primary efficacy measure, the mean change in atrophic lesion area as assessed with FAF, will be assessed at Month 24. In addition to quantifying structural changes of the retina, functional assessments will be performed using scotopic/mesopic microperimetry, as well as standard and low luminance Best-corrected visual acuity (BCVA) evaluations. Total duration of the study for each patient is 30 months following randomization/treatment.

For patients who do not participate in the microperimetry procedure or patients from sites not participating in the microperimetry procedure, there will be only 1 Screening visit, and therefore 13 visits over the study duration.

## 4.1.2 Number of Participants

According to the study protocol, approximately 300 patients (150 per treatment group) will be enrolled in the study at approximately 40 sites. Two hundred forty patients are expected to reach Month 24 for the primary endpoint assessment. The anticipated dropout rate is 20%.

From the patient enrollment monitoring as of September, 2016, total 310 patients were enrolled. Assuming approximately 25% dropout rate based on the survival analysis using Kaplan-Meier estimate, 310 patients will be enough that 240 patients complete the Month 24 visit.

#### 4.2 Study Objectives and Endpoints

Each study objective is presented with corresponding endpoint(s) below:

| Objectives | Endpoints |
|---|---|
| To compare the efficacy of Brimo DDS with<br>Sham in participants with Geographic<br>Atrophy secondary to AMD. | <ul> <li>Primary Endpoint</li> <li>Mean change in atrophic lesion area as assessed with FAF and quantified by the CRC</li> </ul> |
| | <ul> <li>Secondary Endpoint(s)</li> <li>Mean change in low luminance BCVA* as assessed using a 2.0 log unit neutral density filter and the ETDRS visual acuity protocol</li> <li>Mean change in standard BCVA assessed</li> </ul> |
| | <ul> <li>using the ETDRS visual acuity protocol</li> <li>Other Endpoint(s)</li> <li>Mean change in retinal sensitivity threshold as assessed with scotopic/mesopic microperimetry</li> </ul> |
| • To compare the safety of Brimo DDS with Sham treatment procedure in participants with Geographic Atrophy secondary to AMD. | |

<sup>\*</sup> Mean change of low luminance deficit will also be calculated.

#### 5. Statistical Methodology and Study Endpoints

# 5.1 Statistical Methods Planned in the Protocol and Determination of Sample Size

This statistical analysis plan (SAP) will be approved prior to database lock. The SAP expands the statistical section of the protocol and contains a detailed description of methods to analyze data collected in the study. The text portion of the SAP will be included in the CSR report as Appendix 16.1.9.

#### 5.1.1 Statistical and Analytical Plans

Statistical analyses will be conducted using

#### **5.1.1.1** Common Conventions

#### 5.1.1.1.1 Analysis Populations

The analysis populations will consist of participants as defined below:

Table 5-1 Analysis Populations

| Population | Definition | Study Treatment |
|---|---|---|
| Modified Intent-to- All randomized and treated patients with baseline and $\geq 1$ | | As randomized |
| Treat (mITT) postbaseline assessment for geographic atrophy lesion area by | | |
| | FAF, the primary efficacy endpoint. | |
| Safety | All patients who received $\geq 1$ administration of study treatment | As treated |

If a patient is mis-stratified at the randomization, then the patient will be analyzed using the intended stratum in which the patient should belong to.

## **5.1.1.1.2 Study Treatments**

The following treatment groups are defined for this study:

- Brimo DDS 400 μg
- Sham

## 5.1.1.1.3 Statistical Methodology

The methodologies defined below apply as specified to individual endpoints defined in this SAP. When indicated, two-sided 95% confidence intervals and two-sided p-values will be presented. Individual endpoint analyses may specify exceptions (additions or deletions) to these general definitions.

Table 5-2 Statistical Methodology

| Methodology | Description |
|---|---|
| Categorical counts • Number of participants in individual categories ○ Participants with ≥ 1 qualifying event counted once per individual category | |
| Categorical descriptives | <ul> <li>Number and percentage of participants in individual categories</li> <li>○ Participants with ≥ 1 qualifying event counted once per individual category</li> </ul> |
| | <ul> <li>Percentage denominator = N1</li> <li>N1 = participants with non-missing value</li> </ul> |

| Methodology | Description |
|---|---|
| Cumulative | <ul> <li>Cumulative number and percentage of participants in individual categories by</li> </ul> |
| descriptives | visit |
| | <ul> <li>Participants with ≥ 1 qualifying event counted once per individual<br/>category</li> </ul> |
| | <ul> <li>Percentage denominator = number of participants in the population</li> </ul> |
| Continuous | N1, mean, standard deviation (SD), median, minimum, maximum |
| descriptives | • N1 = participants with non-missing value |
| BCVA CFB | BCVA score change from baseline will be classified into the following 5 ordinal |
| categorical<br>change | categories ranked from the best to the worst changes:<br>1) $\geq$ 15 letters improvement; |
| change | <ol> <li>≥ 15 letters improvement;</li> <li>≥ 5 and &lt; 15 letters improvement;</li> </ol> |
| | 3) no change (i.e., change between +5 and -5 letters); |
| | 4) $\geq 5$ and $\leq 15$ letters worsening; |
| | 5) ≥ 15 letters worsening. |
| | • The distribution of the 5 categories at each visit will be summarized by frequency tabulations for each treatment. Treatment comparison will be performed using |
| | Mantel-Haenszel statistics for row mean scores differ using the modified ridit |
| | scores stratified by GA lesion size at screening visit (<= 8 mm <sup>2</sup> , > 8 mm <sup>2</sup> ). |
| CFB MMRM | <ul> <li>Continuous descriptives and standard error (SE) for baseline, postbaseline, and<br/>values at each analysis visit</li> </ul> |
| | <ul> <li>N1 = participants with non-missing values at both baseline and the</li> </ul> |
| | specified postbaseline analysis visit |
| | CFB will be analyzed with a Mixed Model for Repeated Measures (MMRM). |
| | The model includes treatment, study region (North America, Europe, and |
| | Australia), analysis visit, and treatment-by-visit interaction as factors as well as |
| | the baseline value and baseline value-by-analysis visit interaction as covariates. |
| | An unstructured (co)variance structure shared across treatment groups was used |
| | to model the within-patient errors (compound symmetry if convergence fails). |
| | The Kenward-Roger approximation was used to estimate denominator degrees of |
| | freedom and adjust standard errors. Analyses were implemented with SAS PROC |
| | MIXED. The following is the sample SAS codes. |
| | proc mixed; |
| | class subject treatment time region; |
| | model Y = baseline treatment time region |
| | treatment*time baseline*time / ddfm=kr; |
| | repeated time / sub = subject type = un; |
| | lsmeans treatment*time / diff slice=time cl; |
| | estimate 'treatment difference at tx' treatment -1 1 |
| | treatment * time 0 0 0 0 -1 |
| | 0 0 0 0 1/cl; |
| | run; |
| Least squares (LS) means and standard errors | |
| LS mean differences, standard errors, and confidence intervent | |
| | comparing Brimo DDS vs Sham |
| <ul> <li>P-values from contrast t-test comparing Brimo DDS vs Sha</li> <li>N1 = participants with non-missing values at both baseline</li> </ul> | |
| | specified postbaseline analysis visit |
| Nonparametric | Number and percentage of patients in individual categories by treatment group |
| descriptives | <ul> <li>Mantel-Haenszel statistics for row mean scores differ using the modified ridit</li> </ul> |

| Methodology | Description |
|---|---|
| | scores stratified by GA lesion size at screening visit (<= 8 mm <sup>2</sup> , > 8 mm <sup>2</sup> ). |

CFB = change from baseline; AE = Adverse Event

#### **5.1.1.1.4 Missing Data**

For efficacy variables, only observed data will be used.

#### **5.1.1.1.5 Site Pooling**

Region, defined by geographic proximity, will be summarized as North America, Europe and Australia. Sites will be pooled into these three categories.

## 5.1.1.2 Demographics

### 5.1.1.2.1 Analysis Populations

The distribution of participants within the analysis populations will be summarized as follows:

Table 5-3 Analysis Population Summaries

| Population | Variable | Timing | Methodology |
|---|---|---|---|
| mITT, and Safety | Distribution in total and by treatment | _ | Categorical counts |
| populations | group overall and by randomization | | |
| | stratum | | |

## 5.1.1.2.2 Participant Disposition

Participant disposition encompasses the distribution of participants who enter, complete, and discontinue each specified analysis period, along with eCRF-reported discontinuation reasons from each respective analysis period. Participant disposition will be summarized as follows for the All Randomized Population:

Table 5-4 Participant Disposition Summaries

| Parameter | | Variable | Timing | Methodology |
|---|---|---|---|---|
| Dispositions | Numbe | er of participants | Treatment Period <sup>1</sup> | Categorical |
| | 0 | Screened | | descriptives |
| | 0 | Randomized | | |
| | 0 | Treated | | |
| | 0 | Completed | | |
| | 0 | Discontinued | | |
| | <ul> <li>Reason</li> </ul> | s for discontinuation | | |
| | 0 | Adverse Event | | |
| | 0 | Lack of Efficacy | | |
| | 0 | Pregnancy | | |
| | 0 | Lost to Follow-up | | |
| | 0 | Withdrawal by Subject | | |
| | 0 | Protocol Violation | | |
| | 0 | Other | | |
| | | O tilei | | |

<sup>&</sup>lt;sup>1</sup> Treatment period will be defined from baseline to Month 30 or early study exit.

#### **5.1.1.2.3** Protocol Deviations

Protocol deviations will be defined in a separate Protocol Deviation Log, including importance classification. Significant protocol deviations will be summarized as follows:

Table 5-5 Protocol Deviation Summary

| Parameter | Variable | Timing | Methodology |
|---|---|---|---|
| Significant protocol | Distribution in all randomized patients in | | Categorical |
| deviations | total and by treatment group | | descriptives |

#### 5.1.1.2.4 Demographics

Demographics will be summarized in total and by treatment group for the mITT population, as follows:

Table 5-6 Demographic Summaries

| Parameter | Variable | Timing | Methodology |
|---|---|---|---|
| Age | Age (years) relative to informed consent date | Informed consent | Continuous descriptives |
| Age group | <ul><li>&lt; 75 years</li><li>≥ 75 years</li></ul> | Informed consent | Categorical descriptives |
| Sex, race | <ul> <li>eCRF categories</li> <li>Sex</li> <li>Race <ul> <li>White</li> <li>Black</li> <li>Asian</li> <li>Hispanic</li> <li>Other</li> </ul> </li> <li>Race group <ul> <li>White</li> <li>Non-white</li> </ul> </li> </ul> | Screening Visit 1 | Categorical descriptives |

#### **5.1.1.2.5** Baseline Characteristics

Baseline characteristics will be summarized in total and by treatment group for the mITT population as follows:

Table 5-7 Baseline Characteristic and Stratification Factor Summaries

| Parameter | Variable | Timing | Methodology |
|---|---|---|---|
| Baseline characteristics | <ul> <li>Iris Color</li> </ul> | Latest assessment in | Categorical & |
| | o Blue | Screening Period or | Continuous |
| | o Green | Pretreatment Period | descriptives |
| | o Hazel | | |
| | o Brown | | |
| | <ul><li>Other</li></ul> | | |
| | <ul><li>Weight (kg)</li></ul> | | |
| | <ul><li>Height (cm)</li></ul> | | |
| | • BMI $(kg/m^2)$ | | |
| Stratification Factors | Region by Geographic atrophic | Latest assessment in | Categorical |
| | lesion area in study eye as | Screening Period or | descriptives |

| Parameter | Variable | Timing | Methodology |
|---|---|---|---|
| | assessed by FAF at Screening<br>Visit 1 | Pretreatment Period | |
| | <ul> <li>North America</li> <li>≤ 8 mm²</li> <li>&gt; 8 mm²</li> </ul> | | |
| | <ul> <li>Europe</li> <li>≤ 8 mm²</li> <li>&gt; 8 mm²</li> </ul> | | |
| | <ul> <li>Australia</li> <li>≤ 8 mm²</li> <li>&gt; 8 mm²</li> </ul> | | |

#### 5.1.1.2.6 Prior and Concomitant Medications

Medications will be coded using the World Health Organization (WHO) Drug Dictionary, March 2016 or newer. Medication will be listed for the Safety Population defined as follows:

Table 5-8 Prior Medication

| Parameter | Variable | Timing |
|---|---|---|
| Prior medications | <ul> <li>Medications taken ≥ 1 time (see below for time definition) before the study treatment start date, regardless of medication end date. A medication will be defined as a prior medication if it satisfies at least one of the following: <ul> <li>The start date is prior to Day 1, regardless of the stop date;</li> <li>The stop date is prior to or on Day 1, regardless of the start date; or</li> <li>The start date is marked as "&gt; 1 year ago"</li> </ul> </li> </ul> | Screening Period |

**Table 5-9 Concomitent Medication** 

| Parameter | Variable | Timing |
|---|---|---|
| Concomitant medications | <ul> <li>Medications taken ≥ 1 time (see below for time definition) on or after the study treatment start date, regardless of medication start date. A medication will be defined as concomitant if it satisfies at least one of the following:</li> <li>The start date is on or after Day 1, regardless of the stop date;</li> <li>The stop date is after Day 1, regardless of the start date; or</li> <li>The stop date is marked as ongoing.</li> </ul> | Treatment Period |

## **5.1.1.3** Efficacy Analyses

Efficacy analyses will be based on the mITT Population. Baseline for all efficacy endpoints is defined as the last non-missing assessment before the first dose of study treatment.

The following efficacy parameter categorizations are defined:

Table 5-10 Efficacy Assessments

| Assessment | Variable |
|------------|----------|

| Assessment | Variable |
|---|---|
| GA lesion area by FAF | GA lesion area (mm <sup>2</sup> ) as determined by FAF on baseline, Months 6, 12, 18, 24, |
| | and 30 |
| Low luminance BCVA | The number of letters read correctly, quantified using a 2.0 log unit neutral density |
| | filter |
| Standard BCVA | The number of letters read correctly, quantified using the EDTRS visual acuity |
| | protocol. |

#### 5.1.1.3.1 Geographic Atrophy Lesion Area Analyses

Table 5-11 Atrophic Lesion Area Analyses

| Endpoint | Variable | Timing <sup>1</sup> | Methodology |
|---|---|---|---|
| Effective Diameter of GA lesion area (mm) of the study eye by FAF <sup>2</sup> (Primary) | <ul> <li>Means, SDs and other descriptives by visit and treatment group</li> <li>CFB LSMeans, SEs and other descriptives by visit and treatment group</li> <li>Comparison of CFB LS means by visit</li> </ul> | Treatment Period | CFB MMRM |
| Geographic Atrophy<br>Lesion Area (mm²) of<br>the study eye by FAF | <ul> <li>Means, SDs and other descriptives by visit and treatment group</li> <li>CFB LSMeans, SEs and other descriptives by visit and treatment group</li> <li>Comparison of CFB LS means by visit</li> </ul> | Treatment Period | CFB MMRM |

<sup>&</sup>lt;sup>1</sup> Analysis visits defined in Section 6.2.1.

## **5.1.1.3.2** Best Corrected Visual Acuity Analyses

Visual acuity will be recorded on the CRF as the number of letters correctly read. For a given eye, the 4-meter distance (standard) of visual acuity is tested first. If the patient correctly reads at least 20 letters at 4 meters, the visual acuity score will be set as the sum of 30 and the number of letters read correctly. If the patient correctly reads less than 20 letters at 4 meters, the visual acuity is measured again at 1 meter. The visual acuity score will be set to the number of letters read correctly at 1 meter plus the number of letters read correctly at 4 meters.

Table 5-12 Best Corrected Visual Acuity Analyses

| Endpoint | Variable | Timing <sup>1</sup> | Methodology |
|---|---|---|---|
| Low luminance BCVA change from baseline in the study eye (Secondary) | <ul> <li>Descriptive summary of baseline &amp; CFB</li> </ul> | Treatment Period | CFB MMRM |
| Low luminance deficit<br>in the study eye<br>(Secondary) | Descriptive summary of baseline & CFB | Treatment Period | CFB MMRM |
| Standard BCVA change from baseline in the study eye | <ul> <li>Descriptive summary of baseline &amp; CFB</li> </ul> | Treatment Period | CFB MMRM |

<sup>2</sup> Effective diameter (ED) is defined as 2 times square root of GA lesion area divided by  $\pi$  (ED = 2 \*  $\sqrt{GA Area/\pi}$ ).

| Endpoint | Variable | Timing <sup>1</sup> | Methodology |
|---|---|---|---|
| Endpoint (Secondary) Standard BCVA change from baseline in the study eye (Secondary) | <ul> <li>Variable</li> <li>Change in postbaseline BCVA scores from the previous visit will be categorized as <ol> <li>≥ 15 letters improvement;</li> <li>≥ 5 and &lt; 15 letters improvement;</li> <li>no change (i.e., change between +5 and -5 letters);</li> <li>≥ 5 and &lt; 15 letters worsening;</li> </ol> </li> <li>≥ 15 letters worsening</li> </ul> | Timing¹ Treatment Period | BCVA CFB categorical change |

<sup>1</sup> Analysis visits defined in Section 6.2.1.

## **5.1.1.3.3** Exploratory Endpoints and Analyses

Mean change in retinal sensitivity threshold as assessed with scotopic/mesopic microperimetry

The following exploratory efficacy parameter categorizations are defined:

Table 5-13 Exploratory Efficacy Assessments Variable

| Assessment | Variable |
|---|---|
| Retinal sensitivity threshold by scotopic/mesopic microperimetry | The calculated mean retinal sensitivity (dB) from the BEACON test at baseline, Month 6, 12, 18, 24, and 30. |

Retinal sensitivity thresholds in the study eye are measured by MP-1S Microperimetry using a grid with 56 stimulus points at baseline, Month 6, 12, 18, 24 and 30. For each subject at each visit, the mean retinal sensitivity by one of the three neutral density filters (0, 1.0, 2.0) is recorded on the CRF. The mean retinal sensitivity data will be analyzed by each of the three neutral density filters and well as the numeric correction. Correction to the retinal sensitivity values will be conducted as follows: if neutral density filter is 0, then keep the recorded value; if the neutral density filter is 1.0, then add 10dB to the non-zero recorded value; if the neutral density filter is 2.0, then add 20dB to the non-zero recorded value.

Table 5-14 Retinal Sensitivity Threshold Analyses

| Endpoint | Statistics | Timing | Methodology |
|----------|------------|--------|-------------|
|----------|------------|--------|-------------|

| The calculated mean retinal sensitivity (dB) by Neutral Density Filter in the study eye from the BEACON test | Mean, SD and other descriptive statistics by visit and treatment group Change from baseline Mean, SE and other descriptive statistics by visit and treatment group | Treatment Period | Continuous descriptive |
|---|---|---|---|
| 1 | | | |



#### 5.1.1.4.2 Adverse Events

The following adverse event (AE) terms are defined:

Table 5-18 AE Terms

| Term | Variable |
|---|---|
| Treatment | AEs present after the first dose of study treatment or present before the date of the first dose of |
| Emergent | study treatment and increased in severity or became serious after the first dose of study treatment. |
| (TEAE) | |
| Treatment- | Includes TEAEs related to study product or the study procedures as deemed by the study |
| Related | investigator. |
| Ocular | Ocular AEs will be determined based on the OD and OS checked boxes on the AE module of |
| | CRF, and thus are not limited to AEs with SOCs of "Eye." |

Unique participants reporting AEs in the following AE categories will be summarized by treatment group for the Safety Population as follows:

Table 5-19 AE Summaries

| Parameter | Variable | Timing | Methodology |
|---|---|---|---|
| Overall summary | Overall summary only for the following categories: • TEAEs - Ocular - Non-ocular • Treatment-related TEAEs - Ocular - Non-ocular • Serious TEAEs - Ocular - Non-ocular • Deaths • AEs leading to study discontinuation TEAEs by SOC/PT/Severity Treatment Related TEAEs Serious TEAEs AEs leading to study discontinuation | Treatment Period | Categorical descriptives |
| Ocular | TEAEs by SOC/PT | Treatment Period | Categorical |

| Parameter | Variable | Timing | Methodology |
|---|---|---|---|
| | Treatment related TEAEs | | descriptives |
| | Implant/Study Drug-related TEAEs | | _ |
| | Injection Procedure-related TEAEs | | |
| | Applicator-related TEAEs | | |
| Non-ocular | TEAEs by SOC/PT | Treatment Period | Categorical |
| | | | descriptives |

If  $\geq 1$  AE is coded to the same preferred term for the same patient, the patient will be counted only once for that preferred term and strictest causality.

PT and SOC will be ordered by descending frequency by treatment group, ordered from Brimo DDS to Sham, and severity will be ordered by worst severity (maximum severity).







## 5.1.1.5 Subgroup Analyses

Subgroup analysis will be performed based on baseline GA values for the primary endpoint. The subgroup cutoff value will be chosen based on the median of baseline GA size to analyze the data properly.

## 5.1.1.6 Interim Analyses

One interim analysis was conducted when 100% of patients complete the Month-12 visit and 50% of patients complete the Month-18 visit. The study was terminated based on results from the interim analysis.

## **5.1.2 Determination of Sample Size**

Sample size determination was based on previous data or literature (Holz et al, 2010). The following assumptions were made: A GA lesion size of 2.8 mm² for the Sham and 2.1 mm² for the Brimo DDS groups (a 25% reduction from the Sham treatment) and a common SD of 1.65 mm². Under these assumptions, 120 patients will be required in each treatment group to detect the above treatment difference with a power of 90% or greater at the 2-sided t-test with 5%

significance level. With an anticipated dropout rate of 20%, approximately 300 patients will be enrolled such that 240 (120 per group) will complete the Month 24 visit. The sample size calculations are based on the procedure MTTO-1 in nQuery (v6.01).

The sample size assumptions and estimate are summarized as follows:

Table 5-27 Sample Size Assumption

| Parameter | Assumption / Estimate |
|---|---|
| Primary endpoint | Change from baseline in atrophic lesion area in the study eye |
| Mean difference <sup>1</sup> | $0.7 \text{ mm}^2$ |
| $SD^1$ | 1.65 mm <sup>2</sup> |
| α | 5% |
| Sides | 2 |
| Power | 90% |
| Dropout rate | 20% |
| N per group | 150 (120 completing the Month 24 visit) |
| N total | 300 (240 completing the Month 24 visit) |

<sup>&</sup>lt;sup>1</sup> Based on literature (Holz et al, 2010).

## **5.2** Changes in the Conduct of the Study or Planned Analyses

No unplanned analyses were conducted.

#### 5.2.1 Changes in the Conduct of the Study

Prior to database lock, there were no changes in study conduct from what was described in the protocol.

## **5.2.2** Changes to Analyses Prior to Database Lock

According to the study protocol (section 7.1), mITT and safety populations would be analyzed based on the actual treatment that the patient received (as treated). However, the analysis based on mITT population will be conducted based on the treatment to which the patient was randomized (as randomized), and the analysis based on safety population will be based on the actural treatment received. The deviated patients between randomized and actual treatment received will be listed. In addition, analysis based on per-protocol population (PP) will not be performed.

Presence or absence of reticular drusen measured by near-IR (NiR), instead of area of reticular drusen assessed using NiR images, will be analyzed due to the technical difficulties to measure reticular drusen. GA lesion area by FAF in fellow eye was not obtained and will not be analyzed. Medical and ophthalmic history, the atrophic lesion area assessed with SD-OCT examination, and the location of implants and fragments will be not analyzed due to the changed scope of the analyses.

## 6. Data Handling and Analysis Conventions

## **6.1 Study Treatment Conventions**

## 6.1.1 Analysis Days

Treatment days are defined as follows:

Table 6-1 Analysis Day Definitions

| Term | Description |
|---|---|
| Treatment Day | Relative to treatment start date |
| | If analysis date ≥ treatment start date: |
| | <ul> <li>Day = analysis date - treatment start date + 1</li> </ul> |
| | <ul> <li>Day 1 = treatment start date</li> </ul> |
| | If analysis date < treatment start date: |
| | <ul> <li>Day = analysis date – treatment start date</li> </ul> |
| | <ul> <li>Day (-1) = day before treatment start date</li> </ul> |
| | o There is no Day 0 |

## **6.1.2 Missing/Incomplete Treatment End Date**

Not Applicable.





## 6.3 Site Pooling

Region, defined by geographic proximity, will be summarized as North America, Europe and Australia. Sites will be pooled into these three categories.

## **6.4** Missing/Incomplete Date Conventions

Dates may be imputed with year, month, and day values under certain scenarios:

**Table 6-4 Imputation Scenarios** 

| | Complete | | | |
|----------|----------|-------|-----|-----------------|
| Scenario | Year | Month | Day | Imputable |
| 1 | Yes | Yes | Yes | Complete |
| 2 | Yes | Yes | _ | Yes |
| 3 | Yes | _ | Yes | No <sup>1</sup> |
| 4 | Yes | _ | _ | Yes |
| 5 | _ | Yes | Yes | No <sup>1</sup> |
| 6 | _ | Yes | _ | No <sup>1</sup> |
| 7 | | _ | Yes | No <sup>1</sup> |
| 8 | _ | _ | _ | Yes |

| | Complete | | | |
|----------|----------|-------|-----|-----------|
| Scenario | Year | Month | Day | Imputable |

<sup>&</sup>lt;sup>1</sup> Not allowed per database design.

Dates will be imputed initially toward a specified target date for imputable scenarios 2, 4, and 8, and adjusted against the latest reasonable dates. The initial imputed date is determined by the following algorithm:

Table 6-5 Initial Imputed Date Algorithm

| Year (YYYY) of | | Month (MM) of | Incomplete Date | |
|---|---|---|---|---|
| Incomplete Date | Missing | < Target Month | = Target Month | > Target Month |
| Missing | Target Date | _ | _ | _ |
| < Target Year | YYYY-12-31 | _ | YYYY-MM-LD | |
| = Target Year | Target Date | YYYY-MM-LD | Target Date | YYYY-MM-01 |
| > Target Year | YYYY-01-01 | _ | YYYY-MM-01 | _ |

YYYY = year from incomplete date; MM = month from incomplete date; LD = last day of the month.

## 6.4.1 Missing/Incomplete Adverse Event (AE), Start Date

AE start dates will be imputed as the minimum of the following:

- Initial imputed date, where target date = Treatment start date
- Complete end date

## **6.4.2 Missing/Incomplete Medication Start Date**

Medication start dates will be imputed as the minimum of the following:

- Initial imputed date, where target date = Treatment start date -1
- Complete end date

## 6.4.3 Missing/Incomplete AE/Medication End Date

AE and medication end dates will be imputed as the minimum of the following:

- Initial imputed date, where target date = Treatment end date + 30
- Death date

## 6.5 Efficacy Endpoint Conventions

Treatment group will be labeled as follows:

Table 6-6 Treatment Group Label in TFL

| Treatment Group | Presentation |
|----------------------------------------|--------------|
| Brimo DDS <sup>®</sup> contains 400 μg | Brimo DDS |
| brimonidine free base ( | |
| Sham | Sham |

The following conventions will be applied to the TFLs.

Table 6-7 Programming Conventions

| Parameter | Presentation |
|---|---|
| Decimal places | <ul> <li>Summary statistics: For a measure with x decimal places, min and max have x, mean and median have x+1, STD and CI have x+2 decimal places with proper rounding. For ratios such as compliance rate, and daily average scores with</li> <li>x decimal places, min, max, mean and median have x, std and CI have x+1 decimal places with proper rounding.</li> <li>Frequency distribution/incidence rates: % and CI should be rounded to 1 decimal place.</li> </ul> |
| | • P-value: An un-rounded p-value greater than 0.999 should be reported as >0.999. Similarly, an un-rounded p-value less than 0.001 should be reported as <0.001. An un-rounded p-value can be reported as 1.000 only if it is exactly 1.000. Similarly, an unrounded p-value can be reported as 0.000 only if it is exactly 0.000. In presentation, p-values should be rounded to the 3 <sup>rd</sup> decimal place unless it is already determined as >0.999, or <0.001, as discussed earlier. All p-values should be reported with 3 decimal places. Missing p-value will be reported as 'N/A'. |
| P-value approximation | Specify the algorithm of approximation to compute P-values, especially |
| | for non-parametric tests (e.g., Wilcoxon rank sum test, Kruskal-Wallis |
| | test). |

#### 6.6 Safety Endpoint Conventions

#### 6.6.1 Adverse Events

#### 6.6.1.1 Missing Intensity or Relationship

If the investigator is unable to provide the actual values, the following imputations will be applied:

Table 6-8 Missing AE Intensity and Relationship Imputation Algorithms

| Missing Value | Imputation | Timing |
|---------------|------------|---------------------------------------|
| Intensity | Mild | Screening Period, Pretreatment Period |
| | Severe | Treatment Period |
| Relationship | _ | Screening Period, Pretreatment Period |
| | Related | Treatment Period |

## 6.6.2 Repeated or Unscheduled Assessments of Safety Parameters

If end-of-study assessments are repeated or if unscheduled visits occur, the last non-missing post-baseline assessment will be used as the end-of-study assessment for generating summary statistics.

## **6.7 Imputed Value Listing Conventions**

In general, listings will present the actual partial or missing values rather than the imputed values that may be used in endpoint derivation. In instances where imputed values will be presented,

imputed values will be flagged. Actual rules will be fully defined in the table, figure, and data listing specification document.

#### 6.8 Handling Mis-randomization and Mis-stratification

Patients will be randomized by two stratification factors, region (North America, Europe and Australia) and atrophic lesion area ( $\leq 8 \text{ mm2}$  versus > 8 mm2). If a patient is mis-stratified at the randomization, then the patient will be analyzed using the intended stratum in which the patient should have been randomized.

#### 7. References

Holz, FG, Schmidt-Valckenberg S, Fleckenstein M, Jaffe GJ, Hohman T. Lesion characteristics and progression in the natural history of Geographic Atrophy (GAP) Study. Invest Ophthalmol Vis Sci. 2010; 94:a141.

# **ALLERGAN**

## Analysis Plan 190342-038 Final Amend 1

| Date (DD/MMM/YYYY)/Time (PT) | Signed by: | Justification |
|------------------------------|------------|---------------|

#### 1. Title Page

Safety and Efficacy of Brimonidine Posterior Segment Drug Delivery System in Patients with

#### Geographic Atrophy Secondary to Age-Related Macular Degeneration

(BEACON Study: 190342-038)

#### STATISTICAL ANALYSIS PLAN ADDENDUM

#### **SAP** version history:

SAP Version 1.0: February 20, 2017

SAP Version 2.0 Final Amendment: August 3, 2018 SAP Addendum Version 1.0: September 6, 2018

SAP Addendum Version 2.0: March 2019

#### Confidentiality Statement

This document is the property of Allergan, plc. and may not, in full or part, be passed on, reproduced, published, distributed to any person, or submitted to any regulatory authority without the express written permission of Allergan, plc.

#### **SUMMARY OF CHANGES**

The following planned lesion area by SD-OCT analyses will be conducted post-hoc after the DBL:

- 1. Table 14.2-1.7 "Geographic Atrophy Lesion Area (mm2) by SD-OCT: Raw and Change from Baseline"
- 2. Table 14.2-1.8 "Geographic Atrophy Lesion Area (mm2) by SD-OCT: Raw and Change from Baseline; Lesion Area < 4.5 mm2"
- 3. Table 14.2-1.9 "Geographic Atrophy Lesion Area (mm2) by SD-OCT: Raw and Change from Baseline; Lesion Area >= 4.5 mm2"

| Continuous descriptives | <ul> <li>N1, mean, standard deviation (SD), median, minimum, maximum</li> <li>N1 = number of participants with non-missing value</li> </ul> |
|---|---|
| CFB MMRM | <ul> <li>Continuous descriptives for baseline, postbaseline, and CFB values</li> <li>Estimates derived from mixed model for CFB value controlling for factors (treatment group, study region, analysis visit), covariate (baseline GA lesion size as measured by SD-OCT) and interaction (treatment group by analysis visit, treatment group by baseline value). <ul> <li>Least squares (LS) means, standard errors, and 95% confidence intervals for within group change from baseline</li> <li>LS mean differences, standard errors, and confidence intervals vs Placebo</li> <li>P-values from contrast t-test comparing treatment group vs. Placebo</li> <li>N1 = participants with non-missing values at both baseline and the specified postbaseline analysis visit</li> </ul> </li> </ul> |